CLINICAL TRIAL: NCT03493659
Title: The Effects of Standing Tutorials on Problem-Based Learning (PBL) Among Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 00909
Record Dates: First submitted 2018-03-16; First posted 2018-04-10 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2018-03

CONDITIONS: Problem-Based Learning
Keywords: Standing; Sitting; Learning; Problem-Based Learning; Undergraduate

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either a sitting or a standing tutorial, where their learning will be measured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sit-Sit (No Intervention): The participants will sit during the tutorials, and sit during the concept tests given to measure their learning.
- Sit-Stand (Active Comparator): The participants will sit during the tutorials. Intervention: Behavioral: Standing during Concept Test will be administered
  Interventions: Behavioral: Standing during Concept Test
- Stand-Stand (Active Comparator): The participants will stand during the tutorials, and stand during the concept tests given to measure their learning. Intervention: Behavioral: Standing during Concept Test and regular tutorial session will be administered.
  Interventions: Behavioral: Standing during Concept Test and regular tutorial session
- Stand-Sit (Active Comparator): The participants will stand during the tutorials. Intervention: Behavioral: Standing during regular tutorial session will be administered.
  However, participants will sit during the concept tests given to measure their learning.
  Interventions: Behavioral: Standing during regular tutorial session

INTERVENTIONS:
Behavioral: Standing during Concept Test — The participants will stand with a standing desk at an ergonomically correct height during the administration of the Concept Test.
  Arms: Sit-Stand
Behavioral: Standing during regular tutorial session — The participants will stand with a standing desk at an ergonomically correct height during their regular tutorial sessions.
  Arms: Stand-Sit
Behavioral: Standing during Concept Test and regular tutorial session — The participants will stand with a standing desk at an ergonomically correct height during the administration of the Concept Test and during their regular tutorial sessions.
  Arms: Stand-Stand

SUMMARY:
Problem-based learning (PBL) is an education model utilized by Maastricht University and many other universities worldwide. PBL occurs in small, collaborative tutorials, under the facilitation of a tutor. This study explores the effects of standing tutorials, compared against sitting tutorials, on PBL among undergraduate students. A quantitative approach will be taken to objectively measure students' learning, and a qualitative approach will be taken to obtain a deeper understanding of the processes of learning.

It is hypothesized that students in the standing tutorials will be able to recall more academic concepts and link the concepts better than students in the sitting tutorials (H1). Audio-recording of the tutorials will be used to measure the discussions within the tutorials. The transcriptions obtained from the recording will be studied through text analysis. It is hypothesized that students in the standing tutorials will produce more discussions, and therefore a higher word count (H2). It is also hypothesized that the students in the standing tutorials will use more word categories that are conducive to the discussion and learning process (H3).

Through the qualitative approach, the content of the transcriptions will be analysed through a thematic analysis. It is hypothesized that the students in the standing tutorials will produce more learning-oriented interactions (H4).

Two additional factors that would be measured are subsequent physical activity and academic achievement. ActivPAL accelerometers will be used to measure the students' daily activity, to find out if the students' daily activities are affected by the standing tutorials, for example, students may sit more as a result of fatigue from the standing tutorials, or conversely transfer the active behaviour from the standing tutorials to other activities outside the tutorial group.It is hypothesized that standing tutorials do not affect the students' subsequent physical activity, and therefore there will be no significant differences of daily activity between students in the sitting and standing tutorials (H5). With regards to academic achievement, it is hypothesized that the students in the standing tutorials will have higher academic achievements after the course compared to the students in the sitting tutorials (H6).

ELIGIBILITY:
Inclusion Criteria:

* Matriculated undergraduate students of Maastricht University
* Students who have given their consent to participate in this study.
* The course subject is well-established and mandatory for all students within the specific bachelor's programme. A well-established course will be chosen so that clear scoring is possible on the concept tests (explained in the Materials and Analysis sections) that will be administered to the students. The course should be mandatory for all students within the bachelor's programme so as to reduce the selection bias that may otherwise occur if we decide to select tutorial groups that only specific groups of students signed up for. An example of a well-established and mandatory course for students in the Biomedical Sciences bachelor's programme at Maastricht University would include 'Brain, behaviour and movement, 'Human genetics, reproduction and prenatal development' and so on.
* The course coordinators and tutors who are the gatekeepers of the students would have given their permission and cooperation in planning the study into the tutorials.
* The duration of the course would last at least 10 tutorial classes.
* The duration of each tutorial is 2 hours.
* The timing of the tutorial groups will have to be similar to minimize any effects arising due to tests being carried out at different times of the day.
* The course is taught in English.

Exclusion Criteria:

* For the standing tutorials, those who are suffering from musculoskeletal discomfort or pathologies that may prevent or influence movement
* Non-matriculated student of Maastricht University
* Non-matriculated student of the chosen course for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Process of Learning | 1 hour
  The discussions that are carried out during PBL will be audio-recorded and undergo text and thematic analysis
Outcome of Learning | 10 minutes
  Concept Tests will be administered where students list the number of concepts they can recall, and draw a concept map. Both the recalled concepts and the map will be scored independently and combined for a final score.
Academic Achievement | 2 hours
  Grades of Final Exam

SECONDARY OUTCOMES:
Change of Subsequent Physical Activity | 7 days
  Participants' subsequent physical activity will be measured for 10 days, using the ActivPAL accelerometer, to measure whether standing tutorials (compared against sitting tutorials) have an affect on the participants' daily life's physical activity.
Positive and Negative Affect Schedule (PANAS) | 5 minutes
  Participants' overall feelings and emotions are compared between groups in the standing tutorials and sitting tutorials.

OTHER OUTCOMES:
Attendance | Less than 5 minutes (recorded by tutor, as required by the course, even without this intervention study)
  Student attendance across the course are compared to see if attendance is affected by the intervention
Tutor Rating | Less than 5 minutes
  Tutor rating by the students, that the students will give at the end of the course (even without this intervention study)
Search, Preparing and Reporting Phase Questionnaire | 5 minutes
  The questionnaire contains 23 statements, each with a five-point Likert scale describing to what extent the students agreed or disagreed with each statement (1 = 'completely disagree' to 5 = 'completely agree'). Nine statements refer to the theme of "search phase", six statements refer to the theme of "preparing phase", and eight statements refer to the theme of "reporting phase". The aggregate score for each theme will be summed up from the scores on the Likert scale for each statement. Higher scores indicate more effort/preparation for each theme.
Group Interaction Questionnaire | 5 minutes
  This questionnaire is given to tutors to assess the quality of learning-oriented group interactions in PBL. The questionnaire contains 11 statements, each with a five-point Likert scale describing to what extent the tutors agreed or disagreed with each statement (1 = 'completely disagree' to 5 = 'completely agree'). Four statements refer to the theme of "exploratory questions", four statements refer to the theme of "cumulative reasoning", and three statements refer to the theme of "handling conflicts". The aggregate score for each theme will be summed up from the scores on the Likert scale for each statement. Higher scores indicate better discussion quality for each theme.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: December 2019 - depending on the time when summary data are published or otherwise made available.